CLINICAL TRIAL: NCT00541983
Title: A Phase I, Double-blind, Placebo-controlled, Single-dose, Dose-escalation Study of the Safety, Pharmacokinetics, and Preliminary Efficacy of XOMA 052 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Single-dose, Dose-escalation Study of Safety, PK, and Preliminary Efficacy of XOMA 052 in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Pedro Urquilla, MD, XOMA (US) LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X052071
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Type 2; Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: XOMA 052
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XOMA 052 — Subjects in six successive dose groups will receive a single IV infusion (mg/kg) of study drug on Day 0. The total time of the infusion will be 1 hour ± 15 minutes.
  Arms: 1
Drug: Placebo — Subjects in six successive dose groups will receive a single IV infusion (mg/kg) of study drug on Day 0. The total time of the infusion will be 1 hour ± 15 minutes.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK) and preliminary efficacy of XOMA 052 in subjects with active Type 2 Diabetes Mellitus (T2D).

IV administration of XOMA 052 is likely to improve glycemic control in subjects with T2D by blocking certain receptors.

ELIGIBILITY:
Inclusion Criteria:

* American Diabetes Association (ADA) diagnostic criteria for T2D: Fasting blood glucose concentration ≥ 126 mg/dL (≥ 7.0 mmol/L) (must be measured within 28 days prior to Day 0) OR Symptoms of hyperglycemia (e.g., thirst, polyuria, weight loss, visual blurring) AND a casual/random plasma glucose value of ≥ 200 mg/dL (≥ 11.1 mmol/L) (must be measured within 28 days prior to Day 0)
* HbA1c ≥ 7.5% and ≤ 12% (DCCT standard)
* Current T2D of duration > 3 months and ≤ 10 years at Screening
* T2D and other diseases must be stable. Stable disease is defined as disease that is judged stable by the investigator and which did not require a change in medications or dosing level on 4 or more consecutive days or 7 days in total within 28 days prior to Day 0.
* Age ≥ 18 and ≤ 70 at Screening
* Weight ≥ 80 lbs (36.3 kg) and ≤ 325 lbs (147.4 kg)
* BMI ≥ 23 and ≤ 36 kg/m2
* For female subjects of child-bearing age, a negative serum pregnancy test. For subjects with reproductive potential, a willingness to utilize adequate contraception and not become pregnant (or have their partner[s] become pregnant) during the study.
* Agrees not to change diet and exercise regimen during the trial

Exclusion Criteria:

* Use of the following medications: Anti-inflammatory therapy other than aspirin ≤ 100 mg/day; Immunosuppressive treatment; Beta 2 and non-selective adrenergic blockers (Note: selective beta 1 blockers are permitted); Thiazolidinediones; Glucagon-like peptide (GLP) agonists including DPP4 inhibitors
* Change in medication for diabetes within 28 days prior to Day 0, defined as a change in dosing level on 4 or more consecutive days or 7 days in total
* Fasting C-peptide < 400 pM (< 1.20 μg/L)
* Hemoglobin < 8.0 g/dL, WBC < 3.0 × 103/mm3, platelet count < 125 × 103/mm3, creatinine > 1.5 mg/dL, AST/ALT > 2 × ULN, alkaline phosphatase > 2 × ULN
* Positive for GAD65 or IA-2 auto-antibodies
* History or evidence of thyroid abnormalities, including active hyperthyroidism needing medication. Subjects with hypothyroidism will not be excluded if their TSH level has been normal during the 3 months prior to Screening.
* Abnormal T3, T4, thyroglobulin, or TSH levels
* Known HIV antibody, hepatitis B surface antigen, and/or hepatitis C antibody
* History of malignancy within 5 years prior to study entry other than carcinoma in situ of the cervix, or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of tuberculosis, positive PPD test, active atopic disease requiring medication, or asthma
* Infectious disease: CRP > 30 mg/L, fever, or infection requiring treatment with antibiotics within 3 weeks prior to Screening; History of recurrent infection or predisposition to infection; Active leg or foot ulcer
* Immunodeficiency
* Female subjects who are pregnant, planning to become pregnant during the course of the study, or breast-feeding
* History or symptoms of a demyelinating disease
* Clinically significant diabetic macular edema and/or proliferative diabetic retinopathy by history or fundoscopy
* Receipt of a live (attenuated) vaccine within 3 months prior to Screening
* Major surgery within 28 days prior to Day 0
* Participation in an investigational drug or device trial within 30 days prior to Screening
* Use of a therapeutic monoclonal antibody within 90 days prior to Screening
* Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to the study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) at Days 0 and 28. | Day 0 and Day 28

SECONDARY OUTCOMES:
Pharmacokinetic assessments from serum samples collected at time points specified in the protocol. | Dose groups 1 - 5: Day 0 pre-dose through Day 91. Dose group 6: Day 0 pre-dose through Day 364.
Safety assessed by adverse events, vital signs measurements, clinical laboratory assessments, infusion reactions, immune responses to XOMA 052. | Dose groups 1 - 5: Day 0 pre-dose through Day 91. Dose group 6: Day 0 pre-dose through Day 364.
Assessment of inflammatory markers CRP and ESR collected at time points specified in the protocol. | Dose groups 1 - 5: Day 0 pre-dose through Day 91. Dose group 6: Day 0 pre-dose through Day 364.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Urquilla, MD, Study Director — XOMA (US) LLC; Marc Donath, MD, Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Covance Clinical Research (formerly Swiss Pharma Contract), Allschwil
  - Zurich

REFERENCES:
- [Derived] Cavelti-Weder C, Babians-Brunner A, Keller C, Stahel MA, Kurz-Levin M, Zayed H, Solinger AM, Mandrup-Poulsen T, Dinarello CA, Donath MY. Effects of gevokizumab on glycemia and inflammatory markers in type 2 diabetes. Diabetes Care. 2012 Aug;35(8):1654-62. doi: 10.2337/dc11-2219. Epub 2012 Jun 14. PMID 22699287
- [Derived] Cavelti-Weder C, Furrer R, Keller C, Babians-Brunner A, Solinger AM, Gast H, Fontana A, Donath MY, Penner IK. Inhibition of IL-1beta improves fatigue in type 2 diabetes. Diabetes Care. 2011 Oct;34(10):e158. doi: 10.2337/dc11-1196. No abstract available. PMID 21949230